CLINICAL TRIAL: NCT02599415
Title: Studying the Effect of Narrow Band Ultraviolet B Phototherapy on Skin Dendritic (DCs) Cells in Psoriasis Patients
Brief Title: Anti-psoriatic Effect of TL01 Light Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2/044/14
Record Dates: First submitted 2015-03-06; First posted 2015-11-06 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Psoriasis
Keywords: psoriasis patients referred to receive TL01 NB-UVB therapy
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TL01 light treatment (Other): routine treatment with a CE marked device that has been used for this disease for many years
  Interventions: Device: TL01 light treatment

INTERVENTIONS:
Device: TL01 light treatment — Patients received treatment in TL01 cabinet three sessions weekly according to a standard escalating protocol based on minimal erythema dose. Standard dose ranges between 0.55 and 3.13J/cm2.
  Other Names: Waldmnn Gmbh cabinet

SUMMARY:
This is a pilot study to investigate the effect of TL01 narrow band UVB therapy on the resident dermal dendritic cells characterized by expression of CD1c and CD141. These cells were reported to have a role in induction of tolerogenic regulatory T cells and production of IL-10. The investigators proposed to investigate the effect of NB-UVB on these subsets of cells after two weeks of treatment to provide better understanding of the mechanism of action of light treatment.

DETAILED DESCRIPTION:
Six patients with plaque psoriasis were recruited from the phototherapy unit. These patients were referred by their dermatologist to receive narrow-band UVB (TL01) light treatment. Two 6 mm lesional skin punch biopsies were taken at baseline and 2 weeks after commencing the light treatment to study the effect of light on innate immune cells involved in psoriasis pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female psoriasis patients in whom the decision to treat with NB-UVB therapy, as part of their routine clinical care, has been taken by their dermatologist in the age range of 18-70 years.

Exclusion Criteria:

* patients currently on antipsoriatic treatment.

  * Patients with immunosuppressive diseases
  * Patients on immunosuppressive therapies
  * Pregnant or lactating female patients
  * Patients unable to provide a written consentProcedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
determination of the effect of TL01 NB-UVB on numbers of CD1c and CD141 cells | 3 months
  no adverse events recorded after two weeks of TL01 treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No